CLINICAL TRIAL: NCT05805449
Title: The BIO RAMP Trial - BIOlogic Augmented Repair of Complex Anal Fistula Using Acellular Matrix and/or Autologous Platelet-rich Plasma
Brief Title: BIOlogic Augmented Repair of Complex Anal Fistula Using Acellular Matrix and/or Autologous Platelet-rich Plasma
Acronym: BIO RAMP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: CENTER FOR CLINICAL AND TRANSLATIONAL SCIENCES (Unknown)
Responsible Party: Principal Investigator, Jeff Van Eps, MD, Assistant Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HSC-MS-22-0759
Record Dates: First submitted 2023-03-16; First posted 2023-04-10 (Actual); Last update posted 2023-04-10 (Actual); Status verified 2023-04

CONDITIONS: Anal Fistula
MeSH Terms: conditions — Rectal Fistula | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (4):
- Surgery (Sham Comparator): Control patients will receive usual standard of care surgical repair of their complex fistula by The ligation of intersphincteric tract (LIFT) or advancement flap technique without any biologic adjunct.
  Interventions: Procedure: Surgery
- Surgery plus platelet-rich plasma (PRP) (Experimental)
  Interventions: Procedure: Surgery; Other: Platelet-rich plasma (PRP)
- Surgery plus matrix (Experimental)
  Interventions: Procedure: Surgery; Device: Matrix
- Surgery plus PRP plus matrix material (Experimental)
  Interventions: Procedure: Surgery; Other: Platelet-rich plasma (PRP); Device: Matrix

INTERVENTIONS:
Procedure: Surgery — Control patients will receive usual standard of care surgical repair of their complex fistula by LIFT or advancement flap technique without any biologic adjunct.
Other: Platelet-rich plasma (PRP) — Participants will have 40-50cc of peripheral whole blood drawn into a syringe pre-loaded with acid citrate dextrose (ACD) anticoagulant and concentrated PRP harvested by double centrifugation technique using the manufacturer's kit and benchtop centrifuge. This typically yields 5-8cc of PRP that is 18-times more concentrated than baseline.
  Arms: Surgery plus PRP plus matrix material; Surgery plus platelet-rich plasma (PRP)
Device: Matrix — Participants will receive 200g of "paste" matrix and 200g injected at the following sites: the internal opening closure site at level of the sphincter muscle, within the walls of the fistula tract along its length, and within the tissue of an advancement flap particularly at areas of tissue apposition.
  Arms: Surgery plus PRP plus matrix material; Surgery plus matrix

SUMMARY:
The purpose of this study is to compare the clinical effectiveness of augmenting surgical repair of complex anal fistula using autologous PRP and/or micronized acellular porcine urinary bladder matrix (UBM) to usual surgical care alone to prevent fistula recurrence or improve HRQoL, to compare the effects of augmenting surgical repair of complex anal fistula using autologous PRP and/or micronized acellular porcine urinary bladder matrix on early postoperative pain and fecal continence and to assess the cost utility of augmented complex fistula repair relative to usual surgical care

ELIGIBILITY:
Inclusion Criteria:

* complex cryptoglandular transsphincteric anal fistula undergoing surgical repair by LIFT or advancement flap procedure
* English or Spanish speaking and capable of providing informed consent
* Willing to undergo temporary anal seton drainage for requisite time prior to repair
* Participating surgeons will only be eligible if they perform at least 3 repair procedures/year

Exclusion Criteria:

* Unable to reliably complete follow up for 12 months postoperatively
* Primary platelet disorders
* Thrombocytopenia < 150 plt/microliter
* Inability to stop anti-platelet agent > 5 days preoperatively
* Fistula associated with inflammatory bowel disease (IBD), malignancy or pelvic/perineal radiation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2023-02-21 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with fistula recurrence | upto 6 months after surgery
  A fistula recurrence is defined as one or more of the following clinical signs or symptoms after repair: recurrent abscess at the site of repair, chronic drainage or passage of flatus from an external opening of the perineum away from the anal verge, a non-healing external opening that tracks toward anus by probing with fistula probe.
Change in Health-related quality of life (HRQoL) as assessed by the EQ-5D-5L questionnaire | Baseline, 1week post surgery, 2 weeks post surgery, 6 weeks post surgery, 3 months post surgery, 6 months post surgery, and 12 months post surgery.
  This instrument queries subjects on health status related to mobility, self-care, 'usual' activities, pain/discomfort, and anxiety/depression with 5 potential responses ranging from "no problems" to inability to complete the task or extreme levels of pain/depression, correlating to a discrete index score from 1-5, a higher number indicating a worse outcome.The instrument also includes an overall VAS self-rating of health ranging from 0-100, higher number indicating better health.

SECONDARY OUTCOMES:
Number of participants who have post operative pain as assessed by the visual analog scale (VAS) | 14 days after surgery
  This is scored from 0-100, higher number indicating better health
Change in fecal continence as assessed by the Cleveland Clinic Fecal Incontinence (CCFI) scoring tool | Baseline, 2 weeks after surgery,6 weeks after surgery,3 months after surgery,6 months after surgery and 12 months after surgery
  This is a 5 item questionnaire that assesses type of incontinence (solid, liquid, gas, wears pad, lifestyle alteration).
  The frequency with which each type of incontinence occurs is rated on a scale from 0 (never) to 4 (always or to 1/day). The sum of the frequencies is added to yield a total score that can range from 0 to 20, with higher scores indicating higher levels of incontinence.
The relative cost utility of the different treatment strategies as assessed by a questionnaire | 12 months after surgery
  A cost effectiveness analysis (CEA) will be done from the healthcare system perspective assessed as the incremental health system costs (or savings) per fistula recurrence prevented

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey L Van Eps, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No